CLINICAL TRIAL: NCT05364879
Title: The Impact of Prehabilitation Exercise on Frailty and Treatment Outcomes in Ovarian Cancer Patients
Brief Title: Prehabilitation for Ovarian Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NSH Adv Ovarian Cancer Prehab
Record Dates: First submitted 2022-03-30; First posted 2022-05-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Prehabilitation; Exercise; Frailty; Ovarian Cancer; Surgical Complication; Treatment Outcomes; Enhanced Recovery After Surgery
MeSH Terms: conditions — Motor Activity; Frailty; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Circuit-based prehabilitation exercise intervention
  Interventions: Behavioral: Prehabilitation Exercise Intervention

INTERVENTIONS:
Behavioral: Prehabilitation Exercise Intervention — The exercise intervention will consist of light-to-moderate intensity aerobic, resistance, and mobility exercises. These exercises will be performed in a circuit type manner. Participants will perform similar exercises that are modified to meet their individual abilities. Exercise intensity, modifications and substitutions will be determined for each participant based on their medical history, 6 minute walk test results, and baseline frailty scores. Exercise sessions will be performed 3x/wk beginning at 30 min and progressing to 60-min as tolerated for a minimum of four weeks but will continue up until the time of the participants surgery. A hybrid approach will be used for the exercise sessions whereby the participant must attend the first exercise session in person and subsequent sessions will be delivered virtually. Sessions will be overseen by the study Clinical Exercise Physiologist.

SUMMARY:
Individuals with ovarian cancer have very poor survival rates. This is because the cancer is not usually detected until it has reached advanced stages. How long an individual survives also is determined by the cancer treatment they receive. Although there are best treatment practices to improve survival, some women have other conditions that limit treatment options. One such condition seen in as many as 50% of women with advanced ovarian cancer is frailty (an age-related decline in function and health). This is a major concern as doctors will often have to change how the cancer is treated based on the patient being frail. For example, patients living with frailty are less likely to have their full tumor removed during surgery. They are also more likely to have complications with surgery, stay in the hospital longer, and recover less well from surgery overall. Patients living with frailty also are more likely to experience delays in their chemotherapy starting, receive lower doses of chemotherapy and/or receive fewer cycles of chemotherapy. These changes in treatment may decrease how long a patient survives after diagnosis. Thus, research is needed to explore strategies to decrease frailty in patients who require treatment for advanced ovarian cancer. An option gaining more attention is physical exercise (e.g. walking, repeatedly rising from a chair). Exercise performed before surgery, which is called prehabilitation, can improve how well a patient recovers after surgery and increase how long they survive. Research has shown that prehabilitation is very beneficial for patients undergoing surgery for heart disease. However, it is not clear whether prehabilitation works for those with advanced ovarian cancer that are going to have surgery. Therefore, the investigators want to explore how a 4+ week exercise program performed while waiting for surgery for advanced ovarian cancer changes frailty and how a patient recovers after surgery. The investigators will specifically look whether the exercise program: 1) reduces how frail a patient is before surgery; 2) improves how well the patient recovers after surgery; and 3) affects the patient's chemotherapy treatment plan. This study will provide important information about the ability of prehabilitation exercise to improve surgical and treatment outcomes in women with advanced ovarian cancer. Overall, it is believed that exercise has the potential to improve the survival of advanced ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have a confirmed diagnosis of stage III or IV ovarian cancer
* Scheduled to receive cytoreductive surgery as part of their treatment plan
* Must have a minimum of 4-weeks between the time of study enrollment and scheduled surgery
* Be able to attend in-person and/or virtual exercise sessions
* Be fluent in English
* Have oncologist approval

Exclusion Criteria:

* Have already completed surgery
* Unstable cardiac or respiratory disease, injury or any other co-morbid disease that may make it unsafe for participants to exercise
* Significant cognitive impairment (e.g., do not have the capacity to consent, unable to follow exercise instructions)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Frailty Change (baseline to post exercise intervention) | Change from baseline to end of 4+ week intervention (pre-surgery)
  Frailty will be assessed using the Clinical Frailty Scale (CFS). The CFS is a The CFS is a 9-point scale (1 - very fit, through very severely frail to 9 - terminally ill) developed for healthcare professionals to summarize the overall level of fitness/frailty of an individual. The CFS covers domains of mobility, energy, physical activity, and function. The higher the score on the CFS the more frail/less fit an individual is.
Frailty Change (baseline to 1-month post surgery) | Change from baseline to about 1-month post-surgery
  Frailty will be assessed using the Clinical Frailty Scale (CFS). The CFS is a The CFS is a 9-point scale (1 - very fit, through very severely frail to 9 - terminally ill) developed for healthcare professionals to summarize the overall level of fitness/frailty of an individual. The CFS covers domains of mobility, energy, physical activity, and function. The higher the score on the CFS the more frail/less fit an individual is.
Frailty Change (baseline to 3-months post surgery) | Change from baseline to about 3-month post-surgery
  Frailty will be assessed using the Clinical Frailty Scale (CFS). The CFS is a The CFS is a 9-point scale (1 - very fit, through very severely frail to 9 - terminally ill) developed for healthcare professionals to summarize the overall level of fitness/frailty of an individual. The CFS covers domains of mobility, energy, physical activity, and function. The higher the score on the CFS the more frail/less fit an individual is.
Surgical Complexity Score (1-month post surgery) | Surgical complexity will be assessed about 1-month post-surgery.
  Surgical complexity will be assessed based on Enhanced Recovery After Surgery (ERAS) guidelines. Complexity scores will be interpreted as "low" (3 or fewer points), "intermediate" (4-7 points), and "high" (8 or more points).
Post-Surgical Outcomes (1-month post surgery) | Post-surgical outcomes will be assessed about 1-month post-surgery.
  Post-surgical outcomes will be assessed based on Enhanced Recovery After Surgery (ERAS) guidelines. Specific outcomes will include post-op glucose control, analgesia usage, pain, daily weight, early mobilization, and post-operative complications.
Surgical Complications (1-month post surgery) | Surgical complications will be assessed post-surgery about 1-month post-surgery.
  Surgical complications will be assessed based on Enhanced Recovery After Surgery (ERAS) guidelines. Specific outcomes will include length of hospital stay and number of readmissions.
Chemotherapy completion rates (End of Cycle 1) | At the end of cycle 1 (each cycle is 3 weeks). Immediately after the procedure.
  Chemotherapy completion rates will be examined through documentation of total drug dose received, changes in dose, cycle delays, and/or discontinuation of treatment
Chemotherapy completion rates (End of Cycle 2) | At the end of cycle 2 (each cycle is 3 weeks). Immediately after the procedure.
  Chemotherapy completion rates will be examined through documentation of total drug dose received, changes in dose, cycle delays, and/or discontinuation of treatment
Chemotherapy completion rates (End of Cycle 3) | At the end of cycle 3 (each cycle is 3 weeks). Immediately after the procedure.
  Chemotherapy completion rates will be examined through documentation of total drug dose received, changes in dose, cycle delays, and/or discontinuation of treatment
Chemotherapy completion rates (End of Cycle 4) | At the end of cycle 4 (each cycle is 3 weeks). Immediately after the procedure.
  Chemotherapy completion rates will be examined through documentation of total drug dose received, changes in dose, cycle delays, and/or discontinuation of treatment
Chemotherapy completion rates (End of Cycle 5) | At the end of cycle 5 (each cycle is 3 weeks). Immediately after the procedure.
  Chemotherapy completion rates will be examined through documentation of total drug dose received, changes in dose, cycle delays, and/or discontinuation of treatment
Chemotherapy completion rates (End of Cycle 6) | At the end of cycle 6 (each cycle is 3 weeks). Immediately after the procedure.
  Chemotherapy completion rates will be examined through documentation of total drug dose received, changes in dose, cycle delays, and/or discontinuation of treatment

SECONDARY OUTCOMES:
Body Mass Index Change (baseline to post exercise intervention) | Change in BMI from baseline to post 4+ week exercise intervention
  Weight (kg) and height (m) will be used to calculate BMI
Body Mass Index Change (baseline to 1-month post surgery) | Change in BMI from baseline to about 1-month post surgery.
  Weight (kg) and height (m) will be used to calculate BMI
Body Mass Index Change (baseline to 3-months post surgery) | Change in BMI from baseline to about 3-month post surgery.
  Weight (kg) and height (m) will be used to calculate BMI
Aerobic Fitness Change (baseline to post exercise intervention) | Change in aerobic fitness from baseline to post 4+ week intervention (pre-surgery)
  The six-minute walk will be used to calculate aerobic fitness
Aerobic Fitness Change (baseline to 1-month post surgery) | Change in aerobic fitness from baseline to about 1-month post surgery
  The six-minute walk will be used to calculate aerobic fitness
Aerobic Fitness Change (baseline to 3-months post surgery) | Change in aerobic fitness from baseline to about 3-months post surgery
  The six-minute walk will be used to calculate aerobic fitness
Muscular Fitness Change (baseline to post exercise intervention) | Change in muscular fitness will be assessed from baseline to post exercise intervention (pre-surgery)
  Muscular fitness will be assessed using the Canadian Society of Exercise Physiology's Physical Activity Training Protocol (CSEP-PATH) and will include the timed sit-to-stand and grip strength.
Muscular Fitness Change (baseline to about 1-month post surgery) | Change in muscular fitness will be assessed from baseline to 1-month post surgery.
  Muscular fitness will be assessed using the Canadian Society of Exercise Physiology's Physical Activity Training Protocol (CSEP-PATH) and will include the timed sit-to-stand and grip strength.
Muscular Fitness Change (baseline to about 3-months post surgery) | Change in muscular fitness will be assessed from baseline to 3-months post surgery.
  Muscular fitness will be assessed using the Canadian Society of Exercise Physiology's Physical Activity Training Protocol (CSEP-PATH) and will include the timed sit-to-stand and grip strength.
Health-Related Quality of Life Change (baseline to post exercise intervention | Chang in health-related quality of life from baseline to post 4+ week intervention (pre-surgery)
  Health-related quality of life will be assess using the EuroQoL five dimensional questionnaire (EQ-5D-5L). The EQ-5D-DL measures mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; higher scores indicate higher problems
Health-Related Quality of Life Change (baseline to 1-month post surgery) | Chang in health-related quality of life from baseline to about 1-month post surgery
  Health-related quality of life will be assess using the EuroQoL five dimensional questionnaire (EQ-5D-5L). The EQ-5D-DL measures mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; higher scores indicate higher problems
Health-Related Quality of Life Change (baseline to 3-months post surgery) | Change in health-related quality of life from baseline to about 3-months post surgery
  Health-related quality of life will be assess using the EuroQoL five dimensional questionnaire (EQ-5D-5L). The EQ-5D-DL measures mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; higher scores indicate higher problems
Physical, Functional, Emotional, and Social/Family Quality of Life Change (baseline to post exercise intervention) | Change in FACT-O from baseline to post 4+ week intervention (pre-surgery)
  The Functional Assessment of Cancer Therapy for Ovarian Cancer (FACT-O) will be used to measure cancer-specific quality of life; 27-item questionnaire with higher scores indicating higher overall quality of life.
Physical, Functional, Emotional, and Social/Family Quality of Life Change (baseline to 1-month post surgery) | Change in FACT-O from baseline to about 1-month post surgery
  The Functional Assessment of Cancer Therapy for Ovarian Cancer (FACT-O) will be used to measure cancer-specific quality of life; 27-item questionnaire with higher scores indicating higher overall quality of life.
Physical, Functional, Emotional, and Social/Family Quality of Life Change (baseline to 3-months post surgery) | Change in FACT-O from baseline to about 3-months post surgery
  The Functional Assessment of Cancer Therapy for Ovarian Cancer (FACT-O) will be used to measure cancer-specific quality of life; 27-item questionnaire with higher scores indicating higher overall quality of life.

OTHER OUTCOMES:
Study Feasibility - Participant Accrual | Throughout study completion, about 2 years
  Participant accrual calculated as % of patients referred divided by number of patients consented to participation
Study Feasibility - Participant Attrition | Through study completion, about 2 years
  Participant attrition calculated as % of consented patients who complete a minimum of 4 weeks of pre-surgical exercise divided by number who withdraw
Study Feasibility - Participant Adherence | Throughout study completion, about 2 years
  Participant program adherence calculated as % of minimum number of exercise sessions completed (e.g., 3 sessions/week for a minimum of 4 weeks for a total of 12 sessions) divided by total number of available exercise sessions over 12-week intervention
Adverse Events | Throughout study completion, about 2 years
  All exercise-related adverse and serious adverse will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Scott Grandy, PhD, Principal Investigator — Nova Scotia Health
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Laboratory website — http://www.thepaclab.com